CLINICAL TRIAL: NCT06584071
Title: A Phase Ib/II Clinical Trial to Evaluate the Preliminary Efficacy, Safety and Pharmacokinetics of PM8002 Injection Combined With PM1009 Injection in Patients With Locally Advanced or Metastatic Hepatocellular Carcinoma
Brief Title: A Study to Evaluate of PM8002 Combined With PM1009 in Patients With First-line HCC
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biotheus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PM80021009-AB001C-HCC-R
Record Dates: First submitted 2024-08-21; First posted 2024-09-04 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: HCC; Liver Cancer
Keywords: first line; HCC; PM1009; PM8002
MeSH Terms: conditions — Liver Neoplasms | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1- combination treatment (Experimental): Combination regimen：PM8002 combined with PM1009. The drugs are administered on the first day every 3 weeks (Q3W), until disease progression or intolerable toxicity or patient withdrawal or study discontinuation(Whichever occurs first).
  Interventions: Drug: PM8002; Drug: PM1009
- Cohort 2- combination treatment (Experimental): Combination regimen：PM8002 combined with PM1009(low dose). The drugs are administered on the first day every 3 weeks (Q3W), until disease progression or intolerable toxicity or patient withdrawal or study discontinuation(Whichever occurs first).
  Interventions: Drug: PM8002; Drug: PM1009
- Cohort 3- monotherapy (Experimental): PM8002 administered on the first day every 3 weeks (Q3W), until disease progression or intolerable toxicity or patient withdrawal or study discontinuation(Whichever occurs first).
  Interventions: Drug: PM8002
- Cohort 4 (Active Comparator): Combination regimen：atezolizumab combined with bevacizumab. The drugs are administered on the first day every 3 weeks (Q3W), until disease progression or intolerable toxicity or patient withdrawal or study discontinuation(Whichever occurs first).
  Interventions: Drug: atezolizumab; Drug: bevacizumab

INTERVENTIONS:
Drug: PM8002 — PM8002 via IV infusion, Q3W
  Arms: Cohort 1- combination treatment; Cohort 2- combination treatment; Cohort 3- monotherapy
Drug: PM1009 — PM8002 via IV infusion, Q3W
  Arms: Cohort 1- combination treatment; Cohort 2- combination treatment
Drug: atezolizumab — atezolizumab,1200mg, via IV infusion, Q3W
  Arms: Cohort 4
Drug: bevacizumab — bevacizumab,15mg/kg, via IV infusion, Q3W
  Arms: Cohort 4

SUMMARY:
This study to evaluate the preliminary efficacy, safety and pharmacokinetics of PM8002 combined with PM1009 in Patients with first-line Hepatocellular Carcinoma.

DETAILED DESCRIPTION:
The study is divided into two parts. The first part is a phase Ib, single-arm study, which is planned to enroll 3-28 subjects.

The second part is a phase II randomized, parallel-controlled, four-arm, open-label study, which is planned to enroll approximately 120 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in clinical studies;
2. Male or female, aged ≥ 18 years;
3. Pathologically or clinically confirmed (according to AASLD), unresectable locally advanced and/or metastatic HCC;
4. Child-Pugh liver function score ≤7；
5. No prior systemic therapy for locally advanced or metastatic and/or unresectable HCC；
6. At least 1 measurable lesion ；
7. Adequate organ function；
8. ECOG score of 0 to 1；
9. Life expectancy ≥ 12 weeks;

Exclusion Criteria:

1. Pathologically confirmed fibrolamellar HCC, sarcomatoid HCC, cholangiocarcinoma and other components；
2. History of serious allergic diseases；
3. The toxicity of previous anti-tumor therapy has not been alleviated；
4. History of severe cardiovascular diseases within 6 months;
5. Current presence of uncontrolled pleural, pericardial, and peritoneal effusions;
6. History of allogeneic hematopoietic stem cell transplantation or allogeneic organ transplantation;
7. History of alcohol abuse, psychotropic substance abuse or drug abuse;
8. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome;
9. Pregnant or lactating women;
10. Other conditions considered unsuitable for this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | Up to approximately 2 years
  ORR is the proportion of subjects with complete response (CR) or partial response (PR), based on RECIST v1.1.
Optimal dosing regimen of PM8002 in combination with PM1009 | Up to approximately 2 years
  To determine the dosing regimen of PM8002 in combination with PM1009
Treatment related adverse events (TRAEs) | Up to 30 days after last treatment
  The incidence and severity of TRAEs graded according to NCI-CTCAE v5.0

SECONDARY OUTCOMES:
Objective response rate(ORR)(mRECIST) | Up to approximately 2 years
  ORR is the proportion of subjects with complete response (CR) or partial response (PR), based on mRECIST
Disease control rate (DCR) | Up to approximately 2 years
  DCR is defined as the proportion of subjects with complete response (CR), partial response (PR) or stable disease (SD) based on RECIST v1.1 and mRECIST
Duration of response (DOR) | Up to approximately 2 years
  DOR is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first
Progression free survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from the start of treatment until the first documentation of disease progression or death due to any cause, whichever occurs first
Overall survival (OS) | Up to approximately 2 years
  OS is the time from the date of randomization or first dosing date to death due to any cause
Maximum observed concentration [Cmax] | Up to 30 days after last treatment
  To evaluate the Cmax of Combination regimen .
Time to Cmax [Tmax] | Up to 30 days after last treatment
  To evaluate the Tmax of Combination regimen .
Minimum observed concentration [Cmin] | Up to 30 days after last treatment
  To evaluate the Cmin of Combination regimen .
Area under the concentration-time curve [AUC0-last] | Up to 30 days after last treatment
  To evaluate the AUC0-last of Combination regimen .
AUC to the end of the dosing period(AUC0-tau) | Up to 30 days after last treatment
  To evaluate the AUC0-tau of Combination regimen .
Apparent terminal elimination half-life (t1/2) | Up to 30 days after last treatment
  To evaluate the t1/2 of Combination regimen .
Anti-drug antibody (ADA) | Up to 30 days after last treatment
  To evaluate the incidence of ADA to PM8002

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, Principal Investigator — Zhong Shan Hospital, Fudan University

IPD SHARING:
Plan to Share IPD: Yes
The data will be published or presented for publications (poster, abstract,articles or papers) or any presentations
Time Frame: After the trial completed
Access Criteria: NCI is committed to sharing data in accordance with NIH policy.